CLINICAL TRIAL: NCT03599453
Title: Pilot Open Label Clinical Trial Evaluating the Safety and Efficacy of Chemokine Modulation to Enhance the Effectiveness of Pembrolizumab in Patients With Metastatic Triple Negative Breast Cancer
Brief Title: Chemokine Modulation Therapy and Pembrolizumab in Treating Participants With Metastatic Triple-Negative Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: AIM ImmunoTech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 62218
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Triple -Negative Breast Cancer; Estrogen Receptor Negative; HER2/Neu Negative; Anatomic Stage IV Breast Cancer AJCC; Progesterone Receptor Negative
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Biopsy; Celecoxib; Benzenesulfonamides; Introns; Interferon alpha-2; Neurofibromin 2; poly(I).poly(c12,U); Uridine Monophosphate; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (chemokine modulation therapy) (Experimental): Participants undergo pre-treatment biopsy. Participants then undergo chemokine modulation therapy consisting of celecoxib PO BID, recombinant interferon alfa-2b IV over 20 minutes, and rintatolimod IV over 30-60 minutes on days -11 to -9, and -4 to -2. Participants then undergo additional biopsy. Following biopsy and chemokine modulation therapy, participants receive pembrolizumab IV over 30 minutes on day 1. Courses repeat every 3 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy; Procedure: Chemokine Modulation Therapy; Drug: Celecoxib; Biological: Recombinant Interferon Alfa-2b; Drug: Rintatolimod; Biological: Pembrolizumab

INTERVENTIONS:
Procedure: Biopsy — Undergo Biopsy
Procedure: Chemokine Modulation Therapy — Undergo chemokine modulation therapy
Drug: Celecoxib — Given by mouth
  Other Names: Celebrex, YM 177, Benzenesulfonamide
Biological: Recombinant Interferon Alfa-2b — Given intravenously
  Other Names: Alfatronol, Glucoferon, Heberon Alfa, IFN alpha-2B, Interferon alfa 2b, Intron A, recombinant interferon alfa-2b, Recombinant Interferon Alfa-2b, Sch
Drug: Rintatolimod — Given intravenously
  Other Names: 38640-92-5, 616524, Ampligen, Ampligen, Atvogen, Poly(I).Poly(c12,U), Poly(Inosinic Acid) Poly(Cytidylic(12), Uridylic)Acid, RINTATOLIMOD, Rintatolimod
Biological: Pembrolizumab — Given intravenously
  Other Names: Immunoglobulin G4,Keytruda, Lambrolizumab

SUMMARY:
This pilot trial studies how well chemokine modulation therapy works when given prior to pembrolizumab in treating participants with triple-negative breast cancer that has spread to other places in the body. Drugs used in chemokine modulation therapy, such as celecoxib, recombinant interferon alfa-2b, and rintatolimod, work by unleashing or enhancing the cancer immune responses that already exist by either blocking inhibitory molecules or by activating stimulatory molecules. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Giving chemokine modulation therapy before pembrolizumab may work better in treating participants with metastatic triple-negative breast cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

-To evaluate the increase of CD8+ infiltration into tumor microenvironment after pre-treatment CKM regime

SECONDARY OBJECTIVES:

* To evaluate the overall response rate (ORR) to the combination therapy per RECIST v1.1
* To evaluate the efficacy of the chemokine modulation (CKM) in combination with pembrolizumab in patients with metastatic triple negative breast cancer (mTNBC) as compared to historic outcomes of pembrolizumab and other anti-PD1/PD-L1 therapies alone, as determined by secondary measures of efficacy including progression-free survival (PFS), overall survival (OS), and disease control rate (DCR).
* To evaluate the safety profile of CKM regimen given as pre-treatment to pembrolizumab therapy in metastatic breast cancer patients using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

EXPLORATORY OBJECTIVES:

* Examine the immune analysis profile of CKM and pembrolizumab combination.
* Examine the relationship of infiltrating CD4+ and CD8+ T cells and other immune and genetic markers, and their associated PD-1, CD45RA or CD45RO levels.
* Correlate PD-L1 expression within both neoplastic and nonneoplastic stromal elements of the tumor microenvironment to PFS, OS, ORR and adverse events (AEs).
* Correlate Immune Panel results with ORR, PFS, OS and AEs.
* Comparison of response assessment criteria for a prospective analysis

OUTLINE:

Participants undergo pre-treatment biopsy. Participants then undergo chemokine modulation therapy consisting of celecoxib orally (PO) twice daily (BID), recombinant interferon alfa-2b intravenously (IV) over 20 minutes, and rintatolimod IV over 30-60 minutes on days -11 to -9, and -4 to -2. Participants then undergo additional biopsy. Following biopsy and chemokine modulation therapy, participants receive pembrolizumab IV over 30 minutes on day 1. After completion of study treatment, participants are followed up for 90 days and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have pathologically confirmed diagnosis of unresectable or metastatic TNBC with no curative treatment options
* Have been informed of other treatment options
* Patient has lesion that can be biopsied and is willing to undergo the procedure as part of the protocol
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to swallow and retain oral medication
* Have measurable disease per RECIST 1.1 criteria present
* Any line of therapy allowed, radiologically confirmed progression on prior therapy
* No cancer-directed therapy for at least 3 weeks prior to study treatment (bone-directed therapies are allowed)
* Platelets >= 100,000/uL
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1500/uL
* Total bilirubin =< institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Creatinine < ULN OR creatinine clearance >= 50 mL/min per Cockcroft-Gault Equation for patients with creatinine levels greater than ULN
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients currently treated with systemic immunosuppressive agents, including steroids (> than equivalent of 10 mg daily of prednisone), are ineligible until 3 weeks after removal from immunosuppressive treatment (inhaled steroids are allowed)
* Patients with active autoimmune disease or history of transplantation
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Patients with known serious mood disorders (Major depression diagnosis is an exclusion. Other stable mood disorders on stable therapy for > 6 months or not requiring therapy may be allowed after consultation with PI
* Cardiac risk factors including:
* Patients experiencing cardiac event(s) (acute coronary syndrome, myocardial infarction, or ischemia) within 3 months of signing consent
* Patients with a New York Heart Association classification of III or IV
* History of upper gastrointestinal ulceration, upper gastrointestinal bleeding, or upper gastrointestinal perforation within the past 3 years
* Prior allergic reaction or hypersensitivity to nonsteroidal antiinflammatory drugs (NSAIDs) or any drugs administered on protocol
* Prior immunotherapy with anti-PD1/PDL1 therapy for the mTNBC
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drug
* Any patients with a positive Antinuclear Antibodies test will be excluded from study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) as measured by immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) criteria 1.1 | Up to 2 years
  Will be assessed using a Simon two-stage minimax design.

SECONDARY OUTCOMES:
Progression-free survival (PFS) as measured by irRECIST 1.1 criteria | Up to 2 years
  Will be assessed using a Simon two-stage minimax design
Overall survival (OS) as measured by irRECIST 1.1 criteria | Up to 2 years
Disease control rate (DCR) as measured by irRECIST 1.1 criteria | Up to 2 years
  Will be assessed using a Simon two-stage minimax design
Incidence of adverse events graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Up to 2 years
  Adverse events (AEs), serious AEs (SAEs), and toxicities will be summarized by attribution (overall and related/unrelated to treatment) and grade using frequencies and relative frequencies

CONTACTS AND LOCATIONS:
Overall Officials: Shipra Gandhi, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No